CLINICAL TRIAL: NCT06396195
Title: Comparative Evaluation of Clinical Success,Parental and Child Satisfaction of Bioflx Crowns Versus Stainless Steel Crowns as Restorations for Primary Molars: A Randomized Clinical Study
Brief Title: Comparative Evaluation of Bioflx Crowns vs Stainless Steel Crowns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hajar Ashraf, Dr. Hajar Ashraf, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bioflx vs ssc
Record Dates: First submitted 2024-02-15; First posted 2024-05-02 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stainless steel crown (Active Comparator): Tooth preparation will involve using a tapered diamond bur to reduce the occlusal surface by 1-1.5mm. Special attention will be given to ensure a consistent occlusal reduction. Interproximal reduction will be carried out distally using a tapered diamond bur, with the rounding of line angles and achieving a knife-edge finish margin on the proximal surface while avoiding any ledge formation.
  For crown selection, an appropriately sized crown will be chosen based on the mesiodistal width of the prepared tooth, and a trial fit will be performed to prevent blanching before cementation. The crown will be contoured and crimped using crown-contouring and crimping pliers. Afterward, the crown will be smoothed and polished along the entire margin using a rubber wheel. Finally, the crown will be cemented using type 1 Glass ionomer luting cement (Prevest Denpro, India ), and any excess material will be removed with an explorer. The final occlusion will be then verified.
  Interventions: Other: stainless steel crown
- bioflx crown (Active Comparator): Prior to preparation ,selection of crown size will be done by occlusal to occlusal comparison
  - we will maintain cusp inclines and reduce the occlusal by 1-1.5 mm , including the central groove(Tip of football diamond ) buccal and lingual occlusal third of clinical crown will be reduced by football diamond proximal contact will be opened with adjacent teeth by 0.5 mm, creating a feather edge gingival margin ( tip of black stripe diamond ) Roundation all line angles will be done Buccal bulge reduction will be done while maintaining a snug fit Trial fit the crown. Seating direction will be lingual to buccal . Adjustment of the preparation as needed for snug /active fit which should provide some resistance to dislodgement Glass ionomer luting cement (Prevest Denpro, India ) will be used to cement the crown
  Interventions: Other: bioflx crown

INTERVENTIONS:
Other: bioflx crown — The Bioflx crowns are characterized by their flexibility, durability, and adaptability. These crowns are preformed pediatric crowns designed for aesthetics, combining properties found in both stainless steel and zirconia crowns.
  Arms: bioflx crown
Other: stainless steel crown — Stainless steel crowns continue to be considered the "Gold Standard" for posterior full coverage restorations in primary molars
  Other Names: ssc
  Arms: stainless steel crown

SUMMARY:
Comparative Evaluation of Clinical Success,Parental and child Satisfaction of Bioflx Crowns Versus Stainless Steel Crowns as Restorations for Primary Molars: A Randomized Clinical Study

DETAILED DESCRIPTION:
In the field of pediatric dentistry, various materials can be utilized to treat decayed primary teeth, such as composites, glass ionomer cements, or steel crowns. Despite demonstrating acceptable properties, numerous failures are consistently documented, predominantly linked to issues like secondary caries.

Over the course of time, a variety of full-coverage dental restorations have been introduced and integrated into pediatric dental care. Stainless-steel crowns (SSCs) have emerged as the most widely accepted and frequently utilized full-coverage restoration for both primary and permanent teeth in children. Since the 1950s, pediatric dentists globally have favored SSCs due to their exceptional durability, secure cervical fit, cost-effectiveness, and the fact that they require minimal technique sensitivity during the restoration process.

Stainless steel crowns (SSCs) offer robust and dependable full-coverage restorations, remaining in place throughout the lifespan of a primary tooth. However, a notable drawback is the unfavorable metallic appearance, which is disliked by both parents and children. Numerous efforts have been made to develop alternative esthetic substitutes for SSCs, such as composite, polycarbonate, thermoformed plastic, and zirconia.

As the emphasis on esthetics in children has grown, technological progress has successfully brought about the introduction of prefabricated zirconia crowns (ZCs). The adoption of zirconia crowns for primary dentition began in 2008. While zirconia crowns share mechanical properties with metal, they necessitate greater tooth reduction.

The Bioflx crowns are characterized by their flexibility, durability, and adaptability. These crowns are preformed pediatric crowns designed for aesthetics, combining properties found in both stainless steel and zirconia crowns. However, there is a notable absence of scholarly evidence evaluating the properties of Bioflx crowns and their impact on clinical outcomes and parental satisfaction when compared to conventional options. Consequently, this study aims to examine the clinical performance of Bioflx crowns and traditional stainless steel crowns (SSCs) in pediatric patients, with a focus on assessing child and parental satisfaction.

ELIGIBILITY:
Clinical Criteria:

* Children from age 4-7.
* Healthy children .
* Cooperative children and willing for follow-up visits.
* Cariouse Primary Second molars that need pulpotomy and full coverage restorations.

Radiographic criteria:

* Primary molars with two-thirds of the root remaining .
* No widening of PDL space or loss of lamina dura continuity.
* No evidence of internal/external pathologic root resorption.

Exclusion Criteria:

* Uncooperative child .
* Handicapped children either mentally or physically.
* Inability to attend follow-up visits.
* Refuse to participate in the study .
* Tooth with poor prognosis (unrestorable).
* Teeth with root caries .
* Primary teeth with more than half of the root resorbed or presence of periapical pathology seen in the radiograph .

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
crown retention | 12 months
  by tactile examination crown retention scoring (intact or chipped )
parental satisfaction | 12 months
  by a questionnaire-based five-point rating Likert's scale. from (1-5 ) 1= unsatisfied at all to 5 = very satisfied

SECONDARY OUTCOMES:
marginal integrity | 12 months
  crown retention scoring ( open or closed margin )
gingival health | 12 months
  scoring gingival index from (0-3) 0= indicated healthy gingiva to 3 = is severely inflamed gingiva
oral hygiene | 12 months
  by visual clinical examination and score in oral hygiene index (0- 3) 0 =No debris 3 = Soft tissue debris covering more than two third of tooth surface
patient satisfaction | 12 months
  by a questionnaire- based five-point rating Likert's scale. from (1-5 ) counting 1= unsatisfied at all to 5 = very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Adel Abdel Azeem ElBardissy, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aggarwal P, Goyel V, Mathur S, Sachdev V. Effect of Stainless-Steel Crown and Preformed Zirconia Crown on the Periodontal Health of Endodontically Treated Primary Molars Correlating with IL-1beta: An In Vivo Study. J Clin Pediatr Dent. 2022 May 1;46(3):199-203. doi: 10.17796/1053-4625-46.3.5. PMID 35830632
- [Background] Chakraborty, A. et al. (2017) 'Finite element stress analysis of restored primary teeth: A comparative evaluation between stainless steel crowns and preformed Zirconia Crowns', International Journal of Oral Health Sciences, 7(1), p. 10. doi:10.4103/ijohs.ijohs_18_17.
- [Background] Chisini LA, Collares K, Cademartori MG, de Oliveira LJC, Conde MCM, Demarco FF, Correa MB. Restorations in primary teeth: a systematic review on survival and reasons for failures. Int J Paediatr Dent. 2018 Mar;28(2):123-139. doi: 10.1111/ipd.12346. Epub 2018 Jan 10. PMID 29322626
- [Background] Gallagher S, O'Connell BC, O'Connell AC. Assessment of occlusion after placement of stainless steel crowns in children - a pilot study. J Oral Rehabil. 2014 Oct;41(10):730-6. doi: 10.1111/joor.12196. Epub 2014 Jun 10. PMID 24913609
- [Background] Harshitha, A.K. et al. (2021) 'Comparative evaluation on clinical success rate of prefabricated zirconia crowns and stainless steel crowns in primary molars', International Journal of Oral Health Dentistry, 7(3), pp. 180-186. doi:10.18231/j.ijohd.2021.036.
- [Background] Malekzadeh Shafaroudi, A., Nasiri, P. and Nahvi, A. (2021) 'Nickel sensitivity in children due to using stainless steel crowns: A narrative review', Journal of Pediatrics Review, 9(2), pp. 145-152. doi:10.32598/jpr.9.2.870.2.
- [Background] Kilpatrick N, Seow K, Cameron A, et al. Pulp therapy for primary and young permanent teeth. Handbook of Pediatric Dentistry. 2003;2:71-86. [Google Scholar]
- [Background] Mohn M, Frankenberger R, Kramer N. Wear and marginal quality of aesthetic crowns for primary molars. Int J Paediatr Dent. 2022 Mar;32(2):273-283. doi: 10.1111/ipd.12852. Epub 2021 Jul 29. PMID 34138501
- [Background] Nikhil, D.K. et al. (2022) 'Clinical evaluation of Zirconia and stainless-steel crowns in primary molars - a randomized control trial', International Journal of Pedodontic Rehabilitation, 7(2), pp. 30-38. doi:10.56501/intjpedorehab.v7i2.571.
- [Background] O'Connell AC, Kratunova E, Leith R. Posterior preveneered stainless steel crowns: clinical performance after three years. Pediatr Dent. 2014 May-Jun;36(3):254-8. PMID 24960395
- [Background] Patel, M. et al. (2022) 'Clinical evaluation and parental and child satisfaction with restoration of primary teeth using zirconia and stainless steel crowns: A randomized clinical study', Advances in Human Biology, 0(0), p. 0. doi:10.4103/aihb.aihb_43_22.
- [Background] Salman, N. et al. (2021a) 'Parental satisfaction regarding two types of commercial crowns for restoring pulpotomized primary molars', Egyptian Dental Journal, 67(4), pp. 2915-2921. doi:10.21608/edj.2021.93279.1775.
- [Background] Waly AS, Souror YR, Yousief SA, Alqahtani WMS, El-Anwar MI. Pediatric Stainless-Steel Crown Cementation Finite Element Study. Eur J Dent. 2021 Feb;15(1):77-83. doi: 10.1055/s-0040-1715915. Epub 2020 Oct 1. PMID 33003242